CLINICAL TRIAL: NCT00111358
Title: The Effects of a Lifestyle Modification Program (REACH) in Patients With HIV and Metabolic Syndrome
Brief Title: Study of Lifestyle Modification in HIV Lipodystrophy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Steven Grinspoon, MD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 49302-P1 (completed); R01DK049302 (NIH)
Record Dates: First submitted 2005-05-19; First posted 2005-05-20 (Estimated); Last update posted 2011-04-18 (Estimated); Status verified 2011-04

CONDITIONS: HIV; Metabolic Diseases
Keywords: HIV, AIDS, metabolic syndrome
MeSH Terms: conditions — Metabolic Diseases; Acquired Immunodeficiency Syndrome; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lifestyle Modification (Active Comparator): Goals derived from the AACE and NCEP-ATP III guidelines and the Diabetes Prevention Program are as follows: <35% calories from fat, < 7% calories from saturated fat, up to 10% calories from polyunsaturated fat, reduction of trans fatty acid intake, up to 20% calories from monounsaturated fat, and 25-35g of fiber per day. 3 hrs of physical activity/week at moderate intensity, >10,000 steps in daily activity, measured by pedometer. The curriculum is modeled after the Diabetes Prevention Program. Subjects will complete lifestyle sessions in the offices of the Program in Nutritional Metabolism or in the Clinical Research Center at MGH with protocol study staff trained to implement the curriculum.
  Interventions: Behavioral: Lifestyle Modification
- Control (Placebo Comparator)
  Interventions: Other: No lifestyle modification

INTERVENTIONS:
Behavioral: Lifestyle Modification
  Arms: Lifestyle Modification
Other: No lifestyle modification
  Arms: Control

SUMMARY:
This study is designed to determine the effects of an intensive lifestyle modification program in patients with HIV and Metabolic Syndrome. The primary endpoints will be improvement in body composition, specifically waist-to-hip ratio (WHR). The secondary endpoints will include improvement of cardiovascular indices, such as total cholesterol, low-density lipoprotein (LDL), high-density lipoprotein (HDL), and triglyceride cholesterol levels, blood pressure, cardiac enzymes, c-reactive protein (CRP), tissue plasminogen activator (t-PA), plasminogen activator inhibitor (PAI), and insulin and glucose metabolism. We expect that quality of life indices and life skills should also improve with the lifestyle modification program.

DETAILED DESCRIPTION:
This study is designed as a randomized, case-control study of 80 subjects (N=80). Forty subjects will be randomized to the observation group and 40 to the intervention (REACH) group.

After two initial screening visits with medical and nutrition staff for informed consent, determination of eligibility, and evaluation of a 7-day food record, qualifying patients will be seen for a baseline visit. A nutrition questionnaire and bioimpedance analysis (BIA) testing will be done at the first screening visit, and sub-maximal stress testing and other tests with physical therapy will be done at the second screening visit.

At baseline, patients will have an interval history and physical exam, lipodystrophy evaluation by the investigator (objective) and patient (subjective) report, blood tests and body composition.

Nearly identical visits to that at baseline, with the addition of the sub-maximal stress test, and other physical therapy testing, will be repeated at 6 and 12 months. Carotid ultrasound will be repeated at the 6 and 12 month visits. There will also be a short visit at 3 and 9 months to obtain an interval history and physical exam, safety labs, and a 7-day food record for an Intake Report.

At baseline, patients will be randomized to either the observation group or the lifestyle intervention, known as "Reach for Energy, Activity, and Cardiovascular Health" (REACH). Randomization will be stratified for gender and fasting glucose < or >= 110 mg/dL.

Those randomized to observation will receive a one time counseling session with nutrition staff at the baseline visit and monthly, unscripted phone calls from the investigator/co-investigator, and come in for regular study visits at 3, 6, 9, and 12 months, as described above.

Those randomized to REACH will attend one-on-one counseling sessions with a trained dietitian covering the "core-curriculum" that is modeled after the Diabetes Prevention Program (DPP) study 16 week core curriculum intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 and less than or equal to 65 years of age
* HIV+
* Ability and motivation to modify behavior and make lifestyle changes
* 3 out of 5 of the following:

  * Waist circumference greater than 102 cm (40 in) in men and 88 cm (35 in) in women;
  * Triglycerides greater than or equal to 150 mg/dL or current anti-lipolytic drug treatment;
  * High-density lipoprotein (HDL) less than 40 mg/dL in men and 50 mg/dL in women;
  * Blood pressure greater than or equal to 130/85 mmHg or current antihypertensive drug treatment;
  * Fasting glucose greater than or equal to 110 mg/dL.

Exclusion Criteria:

* History of unstable angina, aortic stenosis, uncontrolled hypertension, severe neuropathy, arthritis or other contraindication to exercise
* Requiring pharmacological glucocorticoid therapy (> 7.5mg Prednisone or its equivalent/day)
* Androgen, growth hormone or Megace within 3 months of study initiation. Subjects on a standard dose of testosterone for documented hypogonadism for > 3 months will be allowed to enter the study.
* New anti-retroviral therapy within 1 month of study initiation
* SGPT > 5X normal and/or clinically significant liver disease
* Creatinine > 2.0 mg/dL and/or clinically significant renal disease
* Hemoglobin (Hgb) < 9 g/dL
* Current drug or alcohol abuse
* History of diabetes mellitus or fasting glucose of greater than or equal to 126 mg/dL
* Current therapy with insulin or other diabetic agent
* Pregnant or actively seeking pregnancy
* Breastfeeding
* Inability to comply with intervention due to lack of motivation, time, social, and/or psychological support

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2003-06; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
WHR

SECONDARY OUTCOMES:
total cholesterol
LDL
HDL
triglyceride cholesterol levels
blood pressure
cardiac enzymes
CRP
t-PA
PAI
insulin and glucose metabolism

CONTACTS AND LOCATIONS:
Overall Officials: Steven Grinspoon, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mass General Hospital, Boston, Massachusetts, United States